CLINICAL TRIAL: NCT04799951
Title: A Survey to Assess Knowledge, Attitudes and Practices Amongst Surgeons With Regards to Breast Conservation Surgery and Mastectomy
Brief Title: A Survey to Assess Knowledge, Attitudes & Practices in Surgeons With Regards to Breast Conservation Surgery & Mastectomy
Status: Completed | Type: Observational
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Nita Sukumar Nair, Professor and Surgeon Breast oncology services), Tata Memorial Centre
Other Study IDs: 3212
Record Dates: First submitted 2020-05-26; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Health Personnel Attitude; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast Surgeon: surgeons having experience in and regularly conducting breast conservation surgery and mastectomy surgeries
  Interventions: Other: a survey questionnaire to find knowledge, attitude and practices in treatment of breast cancer.

INTERVENTIONS:
Other: a survey questionnaire to find knowledge, attitude and practices in treatment of breast cancer. — an electronic webbased survey to assess knowledge, attitudes and practices amongst surgeons with regards to breast conservation surgery and mastectomy

SUMMARY:
With increasing evidence the management of breast cancer surgery has seen a paradigm shift towards breast conservation, heralding an era of oncoplastic breast surgery. Despite data supporting BCS(breast conservative surgeries) in suitable patients with early breast cancer, a significant percentage of women in India who would be candidates for BCS still decide to undergo mastectomy. The factors that influence these treatment decisions are complex and involve issues regarding access to health care, concerns for cancer recurrence, and the impact of surgery on body image and sexuality.

Surgeon plays an important role in patient selection for breast conservation based on clinico-pathological characters, explaining to patient regarding mandatory locoregional radiotherapy and regular follow up, helping patient make an informed decision by providing safety and outcome profile as compared to mastectomy. Surgeon's recommendations are considered as important as patient's perception of body image issues, while making the decision. Surgeon's recommendations are usually based on their knowledge and belief regarding patient's disease characteristics and their perceptions regarding patient's socioeconomic capabilities and perceived compliance to prescribed treatment plan.

Hence we are conducting this web based e-survey in surgeons from Private hospitals (breast specific practice) Medical colleges and Regional Cancer Centers (RCC) with an aim to evaluate the to understand knowledge, attitude and practices of primary surgeons regarding breast conservation surgery Vs mastectomy in treatment of breast cancer.

We plan to administer the questionnaire to approximately 100 surgeons, equally distributed within aforementioned sectors.

DETAILED DESCRIPTION:
With increasing evidence the management of breast cancer surgery has seen a paradigm shift towards breast conservation, heralding an era of oncoplastic breast surgery. Despite data supporting BCS in suitable patients with early breast cancer, a significant percentage of women in India who would be candidates for BCS still decide to undergo mastectomy. The factors that influence these treatment decisions are complex and involve issues regarding access to health care, concerns for cancer recurrence, and the impact of surgery on body image and sexuality.

Interestingly, Barron Lerner observed the convergence of the women's liberation movement and the rise of Breast Conservation Surgery as the standard of surgical care in the treatment of early stage disease, implying that the felt need of breast conservation was important in stimulating research into breast conservation. One celebrated example of such demand was, writer Rosamond Babette who refused radical mastectomy when diagnosed with breast cancer in 1971 and sought Bernard Fisher's expertise, who, in that era was offering partial mastectomy for early breast cancer. There is now Level I evidence favoring breast conservation surgery for early breast cancer. Decision of breast conservation surgery or mastectomy for early breast cancer, is based on the clinico-pathological factors, individual factors and physician factors. Each has its influence on the decision; making the decision process complex one.

Age of patient at presentation is important factor and it appears logical that younger patients would prefer breast conservation over mastectomy. Two reviews of the National Cancer Database have demonstrated that on the background of increased numbers of breast conservation younger patients are being treated with mastectomy at higher rates than their older counterparts after adjusting for patient, facility, and tumor characteristics. The subset of women aged ≤ 35 years were twice as likely to undergo mastectomy compared to women aged 61-64 years. These studies also reported similar trends with socioeconomic status, geography, and cancer stage. It is unclear why younger women may be opting for more extensive surgery. This may be due to a concern for locoregional recurrence in younger patients, although more aggressive surgery does not appear to affect breast cancer-specific survival.

Availability of radiation facilities and patients' compliance has been studied in detail with reference to breast conservation. It has been seen that breast conservation rates are higher in tertiary care centers with easy accessibility to radiation facilities and within those patients who stay close by to radiation facilities.

country of training, gender, or number of procedures. These studies suggested female gender, higher case number, training, and individual surgeon practice were associated with increased BCT rates.

TMH Mumbai reports that the proportion of cases undergoing BCS has shown a significant upward trend from 12.6% in 1997 to 70% at present. However at institutes across India BCS rates quoted are less than 30%. Surgeon plays an important role in patient selection for breast conservation based on clinicopathological characters, explaining to patient regarding mandatory locoregional radiotherapy and regular follow up, helping patient make an informed decision by providing safety and outcome profile as compared to mastectomy. Surgeon's recommendations are considered as important as patient's perception of body image issues, while making the decision. Surgeon's recommendations are usually based on their knowledge and belief regarding patient's disease characteristics and their perceptions regarding patient's socioeconomic capabilities and perceived compliance to prescribed treatment plan. We intend to study surgeon's and patient's perspective regarding the decision making, by administering a questionnaire to them.

In an attempt to provide all valid information in easily understandable language and in disambiguous manner various decision making aides have been prepared and studies. In one such study, patients and surgeons were interviewed to identify key factors influencing breast cancer surgery decisions. They were then incorporated into a decision board that could be reviewed at the time of surgical consultation.Randomized trial comparing the decision board to usual care demonstrated that patients who had surgical consultations with the decision board had higher knowledge scores regarding treatment options; less decisional conflict and were more satisfied with the decision-making process. In addition, patients in the decision board group were more likely to undergo BCS (94 vs. 76%, P = 0.03). Recent meta-analysis of studies using decision aids in breast cancer patients, demonstrated that women were 25% more likely to choose BCS over mastectomy if a decision aid was utilized.

Nine studies examined how physician related factors influenced patient's choice of mastectomy versus BCT. The variables reported included comparing individual surgeons' numbers of breast conservations, medical oncology consultation, and specific surgeon demographics such as degree,country of training, gender, or number of procedures. These studies suggested female gender, higher case number, training, and individual surgeon practice were associated with increased BCT rates.

TMH Mumbai reports that the proportion of cases undergoing BCS has shown a significant upward trend from 12.6% in 1997 to 70% at present. However at institutes across India BCS rates quoted are less than 30%. Surgeon plays an important role in patient selection for breast conservation based on clinicopathological characters, explaining to patient regarding mandatory locoregional radiotherapy and regular follow up, helping patient make an informed decision by providing safety and outcome profile as compared to mastectomy. Surgeon's recommendations are considered as important as patient's perception of body image issues, while making the decision. Surgeon's recommendations are usually based on their knowledge and belief regarding patient's disease characteristics and their perceptions regarding patient's socioeconomic capabilities and perceived compliance to prescribed treatment plan.

We intend to study surgeon's perspective regarding the decision making, by administering a questionnaire to them.Aim of this study is to understand knowledge, attitude and practices of primary surgeons regarding breast conservation surgery vs mastectomy in treatment of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* All Surgeon having experience in and working in Breast oncological surgeries

Exclusion Criteria:

* Not Any

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We plan to administer a questionnaire to surgeons working in Private hospital (brest Specific practice) Medical Colleges and Regional cancer centers sectors to gain the relevant information.
  We plan to administer the questionnaire to approximately 100 surgeons.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
knowledge, attitudes and practices of surgeon with regards to breast conservation surgery and mastectomy | 1 year
  to access the knowledge, attitudes and practices of surgeon to study surgeon's and patient's perspective regarding the decision making, by administering a questionnaire to them.

CONTACTS AND LOCATIONS:
Overall Officials: Nita Nair, MCH, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No
As per IEC mandate all data and responses will be kept anonymous hence will not be shared with anyone.

REFERENCES:
- [Background] Bellavance EC, Kesmodel SB. Decision-Making in the Surgical Treatment of Breast Cancer: Factors Influencing Women's Choices for Mastectomy and Breast Conserving Surgery. Front Oncol. 2016 Mar 29;6:74. doi: 10.3389/fonc.2016.00074. eCollection 2016. PMID 27066455
- [Background] NIH consensus conference. Treatment of early-stage breast cancer. JAMA. 1991 Jan 16;265(3):391-5. No abstract available. PMID 1984541
- [Background] Gomez SL, Lichtensztajn D, Kurian AW, Telli ML, Chang ET, Keegan TH, Glaser SL, Clarke CA. Increasing mastectomy rates for early-stage breast cancer? Population-based trends from California. J Clin Oncol. 2010 Apr 1;28(10):e155-7; author reply e158. doi: 10.1200/JCO.2009.26.1032. Epub 2010 Feb 16. No abstract available. PMID 20159812
- [Background] Lautner M, Lin H, Shen Y, Parker C, Kuerer H, Shaitelman S, Babiera G, Bedrosian I. Disparities in the Use of Breast-Conserving Therapy Among Patients With Early-Stage Breast Cancer. JAMA Surg. 2015 Aug;150(8):778-86. doi: 10.1001/jamasurg.2015.1102. PMID 26083835
- [Background] Freedman RA, Virgo KS, Labadie J, He Y, Partridge AH, Keating NL. Receipt of locoregional therapy among young women with breast cancer. Breast Cancer Res Treat. 2012 Oct;135(3):893-906. doi: 10.1007/s10549-012-2156-8. Epub 2012 Sep 5. PMID 22949130
- [Background] Cao JQ, Olson RA, Tyldesley SK. Comparison of recurrence and survival rates after breast-conserving therapy and mastectomy in young women with breast cancer. Curr Oncol. 2013 Dec;20(6):e593-601. doi: 10.3747/co.20.1543. PMID 24311961
- [Background] Ye JC, Yan W, Christos PJ, Nori D, Ravi A. Equivalent Survival With Mastectomy or Breast-conserving Surgery Plus Radiation in Young Women Aged < 40 Years With Early-Stage Breast Cancer: A National Registry-based Stage-by-Stage Comparison. Clin Breast Cancer. 2015 Oct;15(5):390-7. doi: 10.1016/j.clbc.2015.03.012. Epub 2015 Apr 2. PMID 25957740
- [Background] Smith GL, Xu Y, Shih YC, Giordano SH, Smith BD, Hunt KK, Strom EA, Perkins GH, Hortobagyi GN, Buchholz TA. Breast-conserving surgery in older patients with invasive breast cancer: current patterns of treatment across the United States. J Am Coll Surg. 2009 Oct;209(4):425-433.e2. doi: 10.1016/j.jamcollsurg.2009.06.363. Epub 2009 Aug 20. PMID 19801315
- [Background] Chagpar AB, Studts JL, Scoggins CR, Martin RC 2nd, Carlson DJ, Laidley AL, El-Eid SE, McGlothin TQ, Noyes RD, McMasters KM. Factors associated with surgical options for breast carcinoma. Cancer. 2006 Apr 1;106(7):1462-6. doi: 10.1002/cncr.21728. PMID 16470610
- [Background] Morrow M, White J, Moughan J, Owen J, Pajack T, Sylvester J, Wilson JF, Winchester D. Factors predicting the use of breast-conserving therapy in stage I and II breast carcinoma. J Clin Oncol. 2001 Apr 15;19(8):2254-62. doi: 10.1200/JCO.2001.19.8.2254. PMID 11304779
- [Background] Staradub VL, Hsieh YC, Clauson J, Langerman A, Rademaker AW, Morrow M. Factors that influence surgical choices in women with breast carcinoma. Cancer. 2002 Sep 15;95(6):1185-90. doi: 10.1002/cncr.10824. PMID 12216083
- [Background] Churilla TM, Donnelly PE, Leatherman ER, Adonizio CS, Peters CA. Total Mastectomy or Breast Conservation Therapy? How Radiation Oncologist Accessibility Determines Treatment Choice and Quality: A SEER Data-base Analysis. Breast J. 2015 Sep-Oct;21(5):473-80. doi: 10.1111/tbj.12449. Epub 2015 Jul 2. PMID 26133235
- [Background] Nold RJ, Beamer RL, Helmer SD, McBoyle MF. Factors influencing a woman's choice to undergo breast-conserving surgery versus modified radical mastectomy. Am J Surg. 2000 Dec;180(6):413-8. doi: 10.1016/s0002-9610(00)00501-8. PMID 11182389
- [Background] Ganz PA, Schag AC, Lee JJ, Polinsky ML, Tan SJ. Breast conservation versus mastectomy. Is there a difference in psychological adjustment or quality of life in the year after surgery? Cancer. 1992 Apr 1;69(7):1729-38. doi: 10.1002/1097-0142(19920401)69:73.0.co;2-d. PMID 1551058
- [Background] Narendra H, Ray S. Breast conserving surgery for breast cancer: single institutional experience from Southern India. Indian J Cancer. 2011 Oct-Dec;48(4):415-22. doi: 10.4103/0019-509X.92260. PMID 22293254